CLINICAL TRIAL: NCT00000606
Title: National Emphysema Treatment Trial (NETT)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 218
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2009-04

CONDITIONS: Emphysema; Lung Diseases; Lung Diseases, Obstructive; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Emphysema; Lung Diseases; Lung Diseases, Obstructive; Pulmonary Disease, Chronic Obstructive | interventions — Pneumonectomy

INTERVENTIONS:
Procedure: Lung volume reduction surgery

SUMMARY:
To evaluate the long term efficacy, morbidity and mortality associated with medical therapy with lung volume reduction surgery (LVRS) as compared to medical therapy alone and to define patient selection criteria. The trial, conducted in conjunction with a patient registry, is supported by the NHLBI, the Centers for Medicare and Medicaid Services (CMS), and the Agency for Healthcare Research and Quality (AHRQ).

DETAILED DESCRIPTION:
BACKGROUND:

LVRS is intended primarily for those patients whose chronic obstructive pulmonary disease (COPD) is predominantly emphysema. Emphysema is characterized anatomically "by abnormal, persistent enlargement of the airspaces distal to the terminal bronchioles, accompanied by the destruction of the airspace walls and without obvious fibrosis". The loss of the lung architecture leads to compressible peripheral airways that close at higher than normal lung volumes (early airway closure). The increased compliance and the air trapping from early closure leads to hyperinflation of the lung, over distention of the chest wall, a flattened, disadvantaged diaphragm, and ventilation-perfusion mismatch. In the 1950s and 1960s, Dr. Otto Brantigan theorized that surgical excision of multiple wedges of lung would reduce lung volumes, thereby restoring the outward elastic pull on the small airways and reduce airway obstruction. Dr. Brantigan reported that the surgical excision of lung tissue resulted in significant clinical improvement in some cases, but mortality was high. With little objective data and high mortality, the procedure did not gain widespread acceptance.

The experience that diaphragmatic and chest wall function could be restored in emphysema with lung transplantation renewed interest in Dr. Brantigan's work. Improvements in surgical technique have opened the possibility of performing surgical excisions of lung tissue. Recent reports on LVRS have shown improvements in FEV1, FVC, TLC, RV and dyspnea and quality of life assessments.

These reports generated enormous excitement among patients and their doctors. Many centers around the country started performing LVRS with the result that hundreds of patients had the procedure, despite the preliminary nature of the results, the lack of rigorous patient selection criteria and the lack of information on long term outcome. Basic questions remain such as which patient should have the surgery, what protocol should be followed, what physiological tests should be obtained, and what is the long term efficacy of the technique on morbidity, mortality, and quality of life. The mechanisms of benefit and the full cardiopulmonary consequences are unknown.

The concept for the trial originated in the NHLBI Workshop on Evaluation and Research in Lung Volume Reduction Surgery. The initiative was reviewed and approved at the May 1996 National Heart, Lung, and Blood Advisory Council meeting. The Requests for Proposals were released in June, 1996.

DESIGN NARRATIVE:

In the trial, 1218 eligible patients were randomized to receive either medical therapy (610) or medical therapy with LVRS(608). LVRS was performed by median sternotomy or video-assisted thorascopic surgery (VATS). Centers randomized their patients to either a) medical therapy alone versus medical therapy with LVRS by median sternotomy, b) medical therapy alone versus medical therapy with LVRS by VATS, or c) medical therapy alone versus medical therapy with LVRS by median sternotomy versus medical therapy with LVRS by bilateral VATS. Medical therapy included pulmonary rehabilitation and education. Direct comparisons of the two surgical techniques were possible only at the centers that performed both techniques. All arms included intensive pulmonary rehabilitation. The primary endpoints were survival and functional improvement as assessed by maximum workload. Secondary endpoints included morbidity, improvement in pulmonary function, quality of life and performance of activities of daily living. Follow-up exams, including history, physical exams, pulmonary function tests, exercise tests and quality of life assessments, occurred after pre-operative rehabilitation and six and twelve months after surgery and every twelve months thereafter. Recruitment ended July 31, 2002 and follow-up ended in December, 2002.

ELIGIBILITY:
Men and women with end-stage emphysema.

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1996-12; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Piantadosi — Johns Hopkins University

REFERENCES:
- [Background] Rationale and design of the National Emphysema Treatment Trial (NETT): A prospective randomized trial of lung volume reduction surgery. J Thorac Cardiovasc Surg. 1999 Sep;118(3):518-28. doi: 10.1016/s0022-5223(99)70191-1. No abstract available. PMID 10469970
- [Background] Rationale and design of The National Emphysema Treatment Trial: a prospective randomized trial of lung volume reduction surgery. The National Emphysema Treatment Trial Research Group. Chest. 1999 Dec;116(6):1750-61. doi: 10.1378/chest.116.6.1750. PMID 10593802
- [Background] Ramsey SD, Sullivan SD, Kaplan RM, Wood DE, Chiang YP, Wagner JL. Economic analysis of lung volume reduction surgery as part of the National Emphysema Treatment Trial. NETT Research Group. Ann Thorac Surg. 2001 Mar;71(3):995-1002. doi: 10.1016/s0003-4975(00)02283-9. PMID 11269488
- [Background] Drazen JM. Surgery for emphysema--not for everyone. N Engl J Med. 2001 Oct 11;345(15):1126-8. doi: 10.1056/NEJM200110113451511. No abstract available. PMID 11596594
- [Background] National Emphysema Treatment Trial Research Group; Fishman A, Fessler H, Martinez F, McKenna RJ Jr, Naunheim K, Piantadosi S, Weinmann G, Wise R. Patients at high risk of death after lung-volume-reduction surgery. N Engl J Med. 2001 Oct 11;345(15):1075-83. doi: 10.1056/NEJMoa11798. PMID 11596586
- [Background] Rationale and design of the national emphysema treatment trial. A prospective randomized trial of lung volume reduction surgery. The national emphysema treatment trial research group. J Cardiopulm Rehabil. 2000 Jan;20(1):24-36. doi: 10.1097/00008483-200001000-00005. PMID 10680095
- [Background] Scharf SM, Iqbal M, Keller C, Criner G, Lee S, Fessler HE; National Emphysema Treatment Trial (NETT) Group. Hemodynamic characterization of patients with severe emphysema. Am J Respir Crit Care Med. 2002 Aug 1;166(3):314-22. doi: 10.1164/rccm.2107027. PMID 12153963
- [Background] Ramsey SD, Berry K, Etzioni R, Kaplan RM, Sullivan SD, Wood DE; National Emphysema Treatment Trial Research Group. Cost effectiveness of lung-volume-reduction surgery for patients with severe emphysema. N Engl J Med. 2003 May 22;348(21):2092-102. doi: 10.1056/NEJMsa030448. Epub 2003 May 20. PMID 12759480
- [Background] Fishman A, Martinez F, Naunheim K, Piantadosi S, Wise R, Ries A, Weinmann G, Wood DE; National Emphysema Treatment Trial Research Group. A randomized trial comparing lung-volume-reduction surgery with medical therapy for severe emphysema. N Engl J Med. 2003 May 22;348(21):2059-73. doi: 10.1056/NEJMoa030287. Epub 2003 May 20. PMID 12759479
- [Background] Ware JH. The National Emphysema Treatment Trial--how strong is the evidence? N Engl J Med. 2003 May 22;348(21):2055-6. doi: 10.1056/NEJMp030068. Epub 2003 May 20. No abstract available. PMID 12759478
- [Background] Drazen JM, Epstein AM. Guidance concerning surgery for emphysema. N Engl J Med. 2003 May 22;348(21):2134-6. doi: 10.1056/NEJMe030058. Epub 2003 May 20. No abstract available. PMID 12759481
- [Background] Sciurba F, Criner GJ, Lee SM, Mohsenifar Z, Shade D, Slivka W, Wise RA; National Emphysema Treatment Trial Research Group. Six-minute walk distance in chronic obstructive pulmonary disease: reproducibility and effect of walking course layout and length. Am J Respir Crit Care Med. 2003 Jun 1;167(11):1522-7. doi: 10.1164/rccm.200203-166OC. Epub 2003 Feb 20. PMID 12615634
- [Background] McKenna RJ Jr, Benditt JO, DeCamp M, Deschamps C, Kaiser L, Lee SM, Mohsenifar Z, Piantadosi S, Ramsey S, Reilly J, Utz J; National Emphysema Treatment Trial Research Group. Safety and efficacy of median sternotomy versus video-assisted thoracic surgery for lung volume reduction surgery. J Thorac Cardiovasc Surg. 2004 May;127(5):1350-60. doi: 10.1016/j.jtcvs.2003.11.025. PMID 15115992
- [Background] Kaplan RM, Ries AL, Reilly J, Mohsenifar Z; National Emphysema Treatment Trial Research Group. Measurement of health-related quality of life in the national emphysema treatment trial. Chest. 2004 Sep;126(3):781-9. doi: 10.1378/chest.126.3.781. PMID 15364757
- [Derived] Kaplan RM, Sun Q, Ries AL. Quality of well-being outcomes in the National Emphysema Treatment Trial. Chest. 2015 Feb;147(2):377-387. doi: 10.1378/chest.14-0528. PMID 25340383
- [Derived] Kaplan RM, Sun Q, Naunheim KS, Ries AL. Long-term follow-up of high-risk patients in the National Emphysema Treatment Trial. Ann Thorac Surg. 2014 Nov;98(5):1782-9. doi: 10.1016/j.athoracsur.2014.06.031. Epub 2014 Sep 4. PMID 25201722
- [Derived] Argula RG, Strange C, Ramakrishnan V, Goldin J. Baseline regional perfusion impacts exercise response to endobronchial valve therapy in advanced pulmonary emphysema. Chest. 2013 Nov;144(5):1578-1586. doi: 10.1378/chest.12-2826. PMID 23828481
- [Derived] Giardino ND, Curtis JL, Andrei AC, Fan VS, Benditt JO, Lyubkin M, Naunheim K, Criner G, Make B, Wise RA, Murray SK, Fishman AP, Sciurba FC, Liberzon I, Martinez FJ; NETT Research Group. Anxiety is associated with diminished exercise performance and quality of life in severe emphysema: a cross-sectional study. Respir Res. 2010 Mar 9;11(1):29. doi: 10.1186/1465-9921-11-29. PMID 20214820
- [Derived] Hunninghake GM, Cho MH, Tesfaigzi Y, Soto-Quiros ME, Avila L, Lasky-Su J, Stidley C, Melen E, Soderhall C, Hallberg J, Kull I, Kere J, Svartengren M, Pershagen G, Wickman M, Lange C, Demeo DL, Hersh CP, Klanderman BJ, Raby BA, Sparrow D, Shapiro SD, Silverman EK, Litonjua AA, Weiss ST, Celedon JC. MMP12, lung function, and COPD in high-risk populations. N Engl J Med. 2009 Dec 31;361(27):2599-608. doi: 10.1056/NEJMoa0904006. Epub 2009 Dec 16. PMID 20018959
- [Derived] Moy ML, Reilly JJ, Ries AL, Mosenifar Z, Kaplan RM, Lew R, Garshick E; National Emphysema Treatment Trial Research Group. Multivariate models of determinants of health-related quality of life in severe chronic obstructive pulmonary disease. J Rehabil Res Dev. 2009;46(5):643-54. doi: 10.1682/jrrd.2008.09.0127. PMID 19882497
- [Derived] Drummond MB, Blackford AL, Benditt JO, Make BJ, Sciurba FC, McCormack MC, Martinez FJ, Fessler HE, Fishman AP, Wise RA; NETT Investigators. Continuous oxygen use in nonhypoxemic emphysema patients identifies a high-risk subset of patients: retrospective analysis of the National Emphysema Treatment Trial. Chest. 2008 Sep;134(3):497-506. doi: 10.1378/chest.08-0117. Epub 2008 Jul 18. PMID 18641094
- [Derived] Martinez FJ, Han MK, Andrei AC, Wise R, Murray S, Curtis JL, Sternberg A, Criner G, Gay SE, Reilly J, Make B, Ries AL, Sciurba F, Weinmann G, Mosenifar Z, DeCamp M, Fishman AP, Celli BR; National Emphysema Treatment Trial Research Group. Longitudinal change in the BODE index predicts mortality in severe emphysema. Am J Respir Crit Care Med. 2008 Sep 1;178(5):491-9. doi: 10.1164/rccm.200709-1383OC. Epub 2008 Jun 5. PMID 18535255
- [Derived] Snyder ML, Goss CH, Neradilek B, Polissar NL, Mosenifar Z, Wise RA, Fishman AP, Benditt JO; National Emphysema Treatment Trial Research Group. Changes in arterial oxygenation and self-reported oxygen use after lung volume reduction surgery. Am J Respir Crit Care Med. 2008 Aug 15;178(4):339-45. doi: 10.1164/rccm.200712-1826OC. Epub 2008 Jun 5. PMID 18535254
- [Derived] Washko GR, Fan VS, Ramsey SD, Mohsenifar Z, Martinez F, Make BJ, Sciurba FC, Criner GJ, Minai O, Decamp MM, Reilly JJ; National Emphysema Treatment Trial Research Group. The effect of lung volume reduction surgery on chronic obstructive pulmonary disease exacerbations. Am J Respir Crit Care Med. 2008 Jan 15;177(2):164-9. doi: 10.1164/rccm.200708-1194OC. Epub 2007 Oct 25. PMID 17962632
- [Derived] Falk JA, Martin UJ, Scharf S, Criner GJ. Lung elastic recoil does not correlate with pulmonary hemodynamics in severe emphysema. Chest. 2007 Nov;132(5):1476-84. doi: 10.1378/chest.07-0041. Epub 2007 Oct 1. PMID 17908710
- Available data/document: Individual Participant Data Set: NETT — http://biolincc.nhlbi.nih.gov/studies/nett/ — NHLBI provides controlled access to IPD through BioLINCC. Access requires registration, evidence of local IRB approval or certification of exemption from IRB review, and completion of a data use agreement.
- Available data/document: Study Protocol — http://biolincc.nhlbi.nih.gov/studies/nett/
- Available data/document: Study Forms — http://biolincc.nhlbi.nih.gov/studies/nett/